CLINICAL TRIAL: NCT03868228
Title: Pilot Study Assessing the Efficacy of Oxaliplatin Based Pressurised IntraPeritoneal Aerosol Chemotherapy (PIPAC) for the Treatment of Colorectal Peritoneal Metastases
Brief Title: PIPAC for the Treatment of Colorectal Peritoneal Metastases
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: Barts Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 239718; 239718 (Other: IRAS)
Record Dates: First submitted 2019-03-06; First posted 2019-03-11 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Colorectal Neoplasms; Peritoneal Metastases
Keywords: intraperitoneal chemotherapy; PIPAC; pressurised; colorectal cancer; peritoneal metastases
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with PIPAC (Experimental): Patients with colorectal cancer and peritoneal metastases being treated with pressurised intraperitoneal aerosol chemotherapy (PIPAC)
  Interventions: Procedure: Pressurised Intraperitoneal Aerosol Chemotherapy (PIPAC)

INTERVENTIONS:
Procedure: Pressurised Intraperitoneal Aerosol Chemotherapy (PIPAC) — Use of CapnoPen device to aerosolise Oxaliplatin 92mg/m2 chemotherapy 6-8 weekly intervals for intraperitoneal distribution via laparoscopy.
  Other Names: CapnoPen

SUMMARY:
This study would like to assess the efficacy of pressurised intraperitoneal aerosol chemotherapy (PIPAC). This technique delivers chemotherapy directly into the abdomen via a less invasive laparoscopic or 'keyhole' form of surgery. This type of chemotherapy takes the form of an aerosol, similar to the spray of a deodorant for example. The aerosol is administered into the abdomen under pressure, pushing the chemotherapy deeper into the tissues and cancer. This approach does not involve any surgical removal of the cancer.

DETAILED DESCRIPTION:
This study aims to assess the efficacy of a novel intervention for advanced colorectal cancers with peritoneal metastases (i.e. cancers of the colon or rectum which have spread to the internal lining of the abdomen).

Patients diagnosed with peritoneal metastases usually first undertake a period of neoadjuvant systemic chemotherapy prior to consideration of cytoreductive surgery and subsequent hyperthermic intraperitoneal chemotherapy (CRS-HIPEC). If the extent of peritoneal disease remains too significant then CRS-HIPEC is contraindicated.

Not all patients are suitable for cytoreductive surgery and subsequent hyperthermic intraperitoneal chemotherapy (CRS-HIPEC). CRS-HIPEC involves a large cut down the length of the abdomen, surgery to cut away as many of the structures affected by cancer as possible then the bathing the abdomen in heated chemotherapy. This is associated with a considerable risk of complications and a not insignificant risk of death. As such there is a significant unmet need for less invasive effective treatments for patients with extensive colorectal peritoneal metastases (CPM).

This study would like to assess the efficacy of pressurised intraperitoneal aerosol chemotherapy (PIPAC). This technique delivers chemotherapy directly into the abdomen via a less invasive laparoscopic or 'keyhole' form of surgery. This type of chemotherapy takes the form of an aerosol, similar to the spray of a deodorant for example. The aerosol is administered into the abdomen under pressure, pushing the chemotherapy deeper into the tissues and cancer. This approach does not involve any surgical removal of the cancer.

It is an additional treatment to the standard intravenous or oral chemotherapy which would otherwise be administered in isolation for the selected patients. PIPAC would be administered across multiple sessions assuming no disease progression was identified. It can be used in patients undertaking neo-adjuvant systemic chemotherapy before CRS- HIPEC or used throughout treatment for those patients deemed not suitable for CRS-HIPEC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CPM with expected life expectancy of > 6 months.
2. ECOG Scale of Performance Status (PS) scores 0 or 1.
3. 15 mile catchment area to facilitate overseeing systemic chemotherapy administration
4. Concomitant systemic chemotherapy regimens with FOLFIRI, FOLFOX, Mitomycin C & Fluorouracil, Capecitabine (excluding Lonsurf) or without systemic chemotherapy if no systemic options available to patient
5. Neutrophil count on or just before chemotherapy due date of >1.5

Exclusion Criteria:

1. Age <18
2. MDT decision that patient not suitable for PIPAC
3. Decision by Preoperative Assessment Department or Consultant Anaesthetist that patient not fit for general anaesthesia and / or laparoscopy
4. Clinically evident gross ascites
5. Bowel obstruction
6. Bevacizumab as part of systemic chemotherapy regime - time from chemotherapy to surgery would be too long for PIPAC to be feasible
7. Previous bone marrow suppression due to chemotherapy given risk of post-operative neutropenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-02-05 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival assessed by laparoscopy and cross sectional imaging | 2 year follow up or until death

SECONDARY OUTCOMES:
Quality of life assessments - QLQ-C30 questionnaire | Repeated 6-8 weekly before each PIPAC treatment. Trend correlated over period of trial until end of September 2021 and reported thereafter
  European Organisation for Research and Treatment of Cancer (EORTC) Quality of life questionnaire (QLQ-C30 Verison 3). Range 0-100. A high score for a functional scale represents a high/healthy level of functioning whereas a high score for a symptom scale or item represents a high level of symptomatology or problems.
Serious CTCAE adverse events / operative complications related to PIPAC | CTCAE assessed following each PIPAC treatment 6-8 weekly and 90 day period thereafter. Will be fully reported at end of trial September 2021, but any Grades 3, 4 and 5 will be notified contemporaneously
  Common Terminology Criteria for Adverse Events (CTCAE). Grade 1-5 with higher indicating more severe.
PIPAC related safety regulation breaches / adverse events in theatre | Assessed following each PIPAC treatment 6-8 weekly. Ultimately reported at end of trial September 2021

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No